CLINICAL TRIAL: NCT06947590
Title: Efficacy of Mavacamten in Patients With Symptomatic Latent Obstructive Hypertrophic Cardiomyopathy: A Randomized Controlled Trial
Brief Title: Efficacy of Mavacamten in Patients With Symptomatic Latent Obstructive Hypertrophic Cardiomyopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Liu (Other)
Responsible Party: Sponsor-Investigator, Xu Liu, Professor, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MVLOHCM
Record Dates: First submitted 2025-04-20; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: HCM - Hypertrophic Cardiomyopathy; Mavacamten
Keywords: HCM; Mavacamten
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mavacamten Group (Experimental): Patients in this group were treated with Mavacamten, starting at an initial dose of 2.5 mg, administered orally once daily. Subsequent doses were adjusted based on changes in pressure gradients and cardiac function observed during follow-up.
  Interventions: Drug: mavacamten
- Control Group (No Intervention): Patients in this group did not receive Mavacamten treatment and were instead managed with traditional therapies of their choice, such as beta-blockers or calcium channel blockers.

INTERVENTIONS:
Drug: mavacamten — Patients in this group were treated with Mavacamten, starting at an initial dose of 2.5 mg, administered orally once daily. Subsequent doses were adjusted based on changes in pressure gradients and cardiac function observed during follow-up.
  Arms: Mavacamten Group

SUMMARY:
This study aimed to evaluate the efficacy and safety of Mavacamten compared to no treatment in patients with symptomatic latent obstructive hypertrophic cardiomyopathy. The trial was randomized into two groups: Mavacamten group and Non-Mavacamten group. Over the 30-week treatment period, patients underwent a series of assessments at predefined time points, including transthoracic echocardiography, electrocardiogram (ECG), Holter monitoring, NYHA functional classification, Kansas City Cardiomyopathy Questionnaire (KCCQ), and cardiac biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Weight greater than 45 kg.
3. Adequate acoustic windows to allow for accurate transthoracic echocardiograms (TTEs).
4. Diagnosis of latent obstructive hypertrophic cardiomyopathy, in accordance with the current guidelines of the American College of Cardiology Foundation/American Heart Association, European Society of Cardiology, and Chinese Society of Cardiology.
5. Left ventricular ejection fraction (LVEF) ≥55% at rest, confirmed by the echocardiography core laboratory.
6. New York Heart Association (NYHA) Class II or III symptoms at the time of screening.
7. Resting oxygen saturation ≥90% at the time of screening.

Exclusion Criteria:

1. Any acute or severe comorbidities (e.g., severe infections or hematological, renal, metabolic, gastrointestinal, or endocrine dysfunction).
2. Currently using or having used prohibited medications within 14 days prior to screening, such as cytochrome CYP2C19 inhibitors (e.g., omeprazole or esomeprazole) or strong CYP3A4 inhibitors.
3. Life expectancy of less than 1 year.
4. Pregnant or breastfeeding women.
5. History of syncope or sustained ventricular tachyarrhythmia during exercise within the past 6 months.
6. Atrial fibrillation (AF).
7. Patients currently receiving or planning to receive treatment with disopyramide, cibenzoline, ranolazine, or a combination of beta-blockers with verapamil or diltiazem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
The change in peak left ventricular outflow tract (LVOT) gradient | From baseline to week 30.
  The change in peak left ventricular outflow tract (LVOT) gradient, determined by Doppler echocardiography, during exercise or pharmacologic provocation from baseline to week 30.

SECONDARY OUTCOMES:
The proportion of patients with a peak left ventricular outflow tract (LVOT) gradient of less than 30 mmHg. | At week 30.
  The proportion of patients with a peak left ventricular outflow tract (LVOT) gradient of less than 30 mmHg during exercise or pharmacologic provocation at week 30.
The proportion of patients with a peak left ventricular outflow tract (LVOT) gradient of less than 50 mmHg. | At week 30.
  The proportion of patients with a peak left ventricular outflow tract (LVOT) gradient of less than 50 mmHg during exercise or pharmacologic provocation at week 30.
The proportion of patients with at least a one-class improvement in NYHA functional classification. | At week 30.
  The proportion of patients with at least a one-class improvement in NYHA functional classification at week 30.
The change in the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS). | From baseline to week 30.
  The change in the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ-CSS) from baseline to week 30.
The change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels. | From baseline to week 30.
  The change in N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels from baseline to week 30.
The change in high-sensitivity cardiac troponin I (hs-cTnI) levels. | From baseline to week 30.
  The change in high-sensitivity cardiac troponin I (hs-cTnI) levels from baseline to week 30.
Key safety endpoints | From baseline to week 30.
  Key safety endpoints include the incidence and severity of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China